CLINICAL TRIAL: NCT03083483
Title: Utilizing Transcranial Direct Current Stimulation to Enhance Laparoscopic Technical Skills Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00078782
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Results first posted 2018-11-14 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Subjects are randomized into SMA or bilateral M1 tDCS configurations. They are further randomized into active or sham tDCS.
Who Masked: Participant, Investigator
Masking Description: For the tDCS portion of the protocol, the subject and investigator will be blinded to active vs sham. The configuration and order of FLS tasks will be known to both.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Bilateral M1, active tDCS (Experimental): Participants will complete 6 sessions of the FLS peg transfer task over a 7-day time span. Participants randomized to this cohort had tdcs applied over the bilateral M1 areas of the brain by measurement of 20% length of periauricular distance left and right of the vertex. The anode was placed on the left side and the cathode was placed on the right side.
  Interventions: Device: transcranial direct current stimulation (tDCS)
- SMA, active tDCS (Experimental): Participants will complete 6 sessions of the FLS peg transfer task over a 7-day time span. Participants randomized to this cohort had tdcs applied over the supplementary motor area. The cathode was placed 10% of nasion-inion distance above the nasion and 15% of nasion-inion distance anterior to the vertex.
  Interventions: Device: transcranial direct current stimulation (tDCS)
- sham tDCS (Sham Comparator): Participants will complete 6 sessions of the FLS peg transfer task over a 7-day time span. Participants in this group were either randomized into either Bilateral or SMA configurations using the same measurements, but did not receive active stimulation. Half of these subjects will be placed in the SMA configuration and the other half in the bilateral M1 electrode configuration.
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — tDCS will apply a low, direct current for the duration of the study session while the subject is training the specific laparoscopic tasks.
  Other Names: Soterix

SUMMARY:
The purpose of this study is to test the influences of transcranial direct current stimulation (tDCS) on the acquisition of laparoscopic surgical skills. For this purpose, the investigator will compare variants of tDCS in the first of 2 experiments. The second arm of the trial will investigate gaze training in a similar study design. These questions will be evaluated using the validated Fundamentals of Laparoscopic Surgery (FLS) module 1, with the overall goal of developing a surgical training curriculum that achieves expert level skill in an expedited timeframe. This research provides a novel approach to general surgery training that has the potential to reduce the amount of time and repetitions required to achieve expert laparoscopic skills.

DETAILED DESCRIPTION:
Developing expert performance requires assessment of the thought processes underlying performance and continued refinement of skills in order to obtain automaticity and intuition. Therefore, developing expert surgical skill is a process likely to take longer than the length of residency, thereby diminishing the quality of care delivered to patients.

The proposed study will implement novel neuroscience techniques of transcranial direct current stimulation to determine if it has the capacity to accelerate technical surgical skill learning in order to achieve competency and expertise in an earlier timeframe. tDCS is a non-invasive brain stimulation technique that delivers constant, low current stimulation via electrodes placed on the scalp to modify cortical excitability in an area of interest. When applied to the motor cortex, promising data indicates that tDCS-induced changes lead to expedited recovery in stroke patients as well as enhanced learning in healthy individuals.

This technique has never been applied in the training of surgical residents making this project an innovative approach to enhance skill development.

Experiment 1: Determine if tDCS can accelerate the learning of laparoscopic skills.

In this experiment the investigators will compare behavioral learning curves from FLS modules 1 and 5 in three cohorts who undergo either active tDCS to the bilateral motor cortex (bilateral configuration), active tDCS to the supplementary motor cortex (SMA configuration), or sham tDCS (half in each configuration). This will be tested in groups of 20 participants who train for 40-minutes in each of 6 sessions that occur within 3 weeks. The investigators hypothesize that both active bilateral and SMA tDCS will lead to faster skill acquisition as measured by trials required to gain proficient completion scores (calculated as time plus errors), relative to sham.

The investigators hypothesize that both bilateral and vertex tDCS will lead to faster skill acquisition, with bilateral greater than vertex as measured by trials required to gain proficient module completion scores, relative to the group of participants who practice without active tDCS.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years, healthy male and female
2. Negative urine pregnancy test for female participants
3. Willing and able to provide informed consent
4. Able to follow study procedures

Exclusion Criteria:

1. Indwelling metallic implants
2. Neurological or psychiatric medical history
3. Drug or alcohol abuse
4. Current or prior brain tumor
5. Current or prior seizures
6. Neuroactive medications
7. Current pregnancy
8. Damage, rash, or skin lesion in area of electrode placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morgan L Cox, MD, Principal Investigator — Duke University; Greg Appelbaum, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cox ML, Deng ZD, Palmer H, Watts A, Beynel L, Young JR, Lisanby SH, Migaly J, Appelbaum LG. Utilizing transcranial direct current stimulation to enhance laparoscopic technical skills training: A randomized controlled trial. Brain Stimul. 2020 May-Jun;13(3):863-872. doi: 10.1016/j.brs.2020.03.009. Epub 2020 Mar 19. PMID 32289719

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period ran from 5/1/17 to 12/20/17. Subjects were recruited off of the Duke University Behavioral Research Lab Sessions Scheduling Website for undergraduate and graduate students, Duke School of Medicine students in the Trent Semans Center and Duke South Clinics, and Duke Pre-Medical undergraduate students.
Pre-assignment Details: 2 participants were screen failures
Groups:
- Sham tDCS: Participants will complete 6 sessions of the FLS peg transfer task over a 7-day time span. Participants in this group were either randomized into either Bilateral or SMA configurations using the same measurements, but did not receive active stimulation.
Period: Overall Study
Arm/Group | Bilateral M1, Active tDCS | SMA, Active tDCS | Sham tDCS
Started | 24 | 22 | 23
Completed | 20 | 20 | 20
Not Completed | 4 | 2 | 3
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — technological issues | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Bilateral M1, Active tDCS | SMA, Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (5.2) | 23.5 (5.4) | 22.7 (3.7) | 22.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 14 | 42
  Male | 8 | 4 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 7
  Not Hispanic or Latino | 18 | 17 | 18 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 9 | 6 | 5 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 3 | 2 | 4 | 9
  White | 6 | 10 | 8 | 24
  More than one race | 1 | 2 | 1 | 4
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Time to Completion
Description: Completion time for each repetition of Fundamentals of Laparoscopic Surgery (FLS) task 1 in post-test (1 single repetition of the task that was timed after all training was completed)
Time Frame: 7 days
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: seconds to completion in post test
Arm/Group | Bilateral M1, Active tDCS | SMA, Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20 | 20
seconds to completion in post test | 55.3 (15.4) | 54.5 (13.1) | 59.5 (18.3)

2. Secondary Outcome: Number of Tasks Completed
Description: The number of completed tasks will be calculated during retrospective review of recorded video through study completion. The six training sessions for data collection will be completed within a 7-day span.
Time Frame: 7 days
Population: In performing the study, only FLS task 1 was performed and evaluated. Therefore, no data was collected or analyzed on multiple tasks.
Arm/Group | Bilateral M1, Active tDCS | SMA, Active tDCS | Sham tDCS
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Errors
Description: The number of errors (as defined by FLS) during completion of tasks will be recorded and transitioned into a time addition. This will be collected for every repetition performed during the 6 separate training sessions within a 7-day period. These errors will be defined and retrospective review of recorded video through study completion.
Time Frame: 7 days
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Bilateral M1, Active tDCS | SMA, Active tDCS | Sham tDCS
Number analyzed (Participants) | 20 | 20 | 20
errors
  Drops out of view- session 1 | 1.3 (1.6) | 1.4 (1.6) | 1.2 (1.2)
  Drops out of view- Session 2 | 1.5 (1.4) | 1.6 (1.7) | 1.5 (1.7)
  Drops out of view- Session 3 | 1.2 (1.2) | 1.8 (1.3) | 1.3 (1.7)
  Drops out of view- Session 4 | 1.7 (2.0) | 0.8 (0.9) | 1.2 (1.3)
  Drops out of view- Session 5 | 1.3 (1.4) | 1.8 (1.9) | 1.7 (0.7)
  Drops out of view- Session 6 | 1.0 (1.1) | 1.2 (1.4) | 1.0 (1.7)
  Improper Transfers- Session 1 | 3.8 (12.9) | 3.1 (6.6) | 2.2 (3.3)
  Improper Transfers- Session 2 | 4.8 (14) | 1.5 (2.4) | 1.2 (2.2)
  Improper Transfers- Session 3 | 1.1 (2.1) | 1.0 (1.6) | 0.7 (1.4)
  Improper Transfers- Session 4 | 0.7 (1.3) | 1.0 (1.5) | 1.4 (3.0)
  Improper Transfers- Session 5 | 0.8 (2.6) | 0.7 (0.9) | 1.0 (2.4)
  Improper Transfers- Session 6 | 2.0 (5.8) | 0.7 (0.9) | 1.1 (2.2)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Bilateral M1, Active tDCS | SMA, Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 1/21 | 1/21 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilateral M1, Active tDCS (N=21) | SMA, Active tDCS (N=21) | Sham tDCS (N=21)
Lightheadedness (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) — tDCS stimulation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT03083483/Prot_SAP_000.pdf